CLINICAL TRIAL: NCT05932290
Title: Comparative Effectiveness of Elranatamab (PF-06863135) in Clinical Study C1071003 Versus Standard of Care (SOC) in Real-World (RW) External Control Arms in Patients With Triple-Class Refractory (TCR) Multiple Myeloma (MM)
Brief Title: A Study to Learn About the Effectiveness of the Medicine Called Elranatamab in People With Relapsed Refractory Multiple Myeloma
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C1071031
Record Dates: First submitted 2023-06-14; First posted 2023-07-06 (Actual); Results first posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Multiple Myeloma
Keywords: Myeloma; Multiple Myeloma; relapsed Multiple Myeloma; refractory Multiple Myeloma; PF-06863135; BCMA; bispecific; bispecific antibody; BCMA-CD3 bispecific; Elranatamab; MagnetisMM-3
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Elranatamab: Patients treated with elranatamab from the MagnetisMM-3 trial
  Interventions: Drug: Elranatamab
- Standard of care: Patients treated with standard-of-care therapies from real-world data sources
  Interventions: Drug: Standard of care

INTERVENTIONS:
Drug: Elranatamab — BCMA-CD3 bispecific antibody
  Groups: Elranatamab
Drug: Standard of care — Standard of care
  Groups: Standard of care

SUMMARY:
This study is to understand how well elranatamab (PF-06863135) may be used for relapsed refractory multiple myeloma (RRMM). Sometimes MM might improve at first, but then gets resistant to the treatment and starts growing again (known as relapsed refractory). This study medicine will be compared with standard-of-care (SOC) therapies used in real-world clinical practice. For people receiving elranatamab, the investigators will use data from the phase 2 clinical trial (MagnetisMM-3). The investigators will also use data from multiple real-world sources, representing the SOC in clinical practice. This study does not seek any participants for enrollment. The investigators will compare the experiences of people receiving elranatamab to people receiving SOC therapies. This way, it will help the investigators to know how well elranatamab can be used for RRMM treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older at index date
* Diagnosis of MM
* Measurable disease according to IMWG criteria
* ECOG performance status ≤2
* Refractory to at least 1 proteasome inhibitor, 1 immunomodulatory drug, and 1 anti-CD38 treatment (ie, triple-class refractory [TCR])
* At least 1 treatment following their TCR eligibility

Exclusion Criteria:

* Acute plasma cell leukemia
* Amyloidosis
* Smoldering MM
* Stem cell transplant within 12 weeks of index or active graft versus host disease (GVHD)
* Active malignancy within 3 years before index, except for basal cell or squamous cell skin cancer or carcinoma in situ
* Administration with an investigational drug within 30 days prior to index

Min Age: 18 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with elranatamab will come from the MagnetisMM-3 trial. Patients treated with the standard-of-care therapies will come from real-world data sources.
Sampling Method: Non-Probability Sample
Enrollment: 514 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Costa LJ, LeBlanc TW, Tesch H, Sonneveld P, Kyle RP, Sinyavskaya L, Hlavacek P, Meche A, Ren J, Schepart A, Aydin D, Nador G, DiBonaventura MD. Elranatamab efficacy in MagnetisMM-3 compared with real-world control arms in triple-class refractory multiple myeloma. Future Oncol. 2024;20(17):1175-1189. doi: 10.2217/fon-2023-0995. Epub 2024 Feb 28. PMID 38415370
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C1071031

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This retrospective cohort study used participant level data from study C1071003 (NCT04649359), and external control arms identified from real world data (RWD) sources.
Groups:
- C1071003 Cohort A: Eligible participants with triple-class refractory multiple myeloma (TCR MM), who were B-cell maturation antigen (BCMA) naïve, who were enrolled between 2 February 2021 to 07 January 2022 and who were treated with elranatamab in study C1071003 were included.
- RWD: COTA: Eligible participants with TCR MM who were treated with standard of care (SOC) therapies in real world clinical practice setting, identified from COTA database were included. This arm served as external control arm.
- RWD: Flatiron Health: Eligible participants with TCR MM who were treated with SOC therapies in real world clinical practice setting, identified from Flatiron Health database were included. This arm served as external control arm.
Period: Overall Study
Arm/Group | C1071003 Cohort A | RWD: COTA | RWD: Flatiron Health
Started | 123 | 239 | 152
Completed | 123 | 239 | 152
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Eligible participants whose data was included for observation in this study.
Groups:
- C1071003 Cohort A: Eligible participants with TCR MM, who were BCMA naïve, who were enrolled between 2 February 2021 to 07 January 2022 and who were treated with elranatamab in study C1071003 were included.
- RWD: COTA: Eligible participants with TCR MM who were treated with SOC therapies in real world clinical practice setting, identified from COTA database were included. This arm served as external control arm.
- Total: Total of all reporting groups
Arm/Group | C1071003 Cohort A | RWD: COTA | RWD: Flatiron Health | Total
Number analyzed (Participants) | 123 | 239 | 152 | 514
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.1 (9.4) | 68.0 (9.4) | 69.5 (10.0) | 68.2 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 109 | 72 | 236
  Male | 68 | 130 | 80 | 278
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 72 | 175 | 102 | 349
  Non-white | 51 | 64 | 50 | 165

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS): Study C1071003 Cohort A Versus RWD COTA Cohort- Using Unweighted Analysis
Description: PFS: a) C1071003 Cohort A: time from the date of the first dose until confirmed progressive disease (PD) per IMWG criteria or death due to any cause, whichever occurred first; b) RWD COTA: time from initiation of the first line after participant identified as having TCR MM to either the date of progression or death due to any cause, whichever occurred first. IMWG criteria for progression: an increase of >=25% (Percent) from the lowest response value in any 1 or more of the criteria: serum protein electrophoresis (SPEP) with an absolute increase >0.5 gram/deciliter (g/dL); 24-hour(h) urine protein electrophoresis (UPEP) with an absolute increase >200 microgram (mg)/24 h; in participants without measurable serum and urine M-protein, the absolute increase of >10 mg/dL in the difference between involved and uninvolved free light chain (FLC) levels; or an absolute bone marrow plasma cell >10%. Retrospective data was retrieved and observed in the current study for approximately 1.5 months.
Time Frame: C1071003:First dose to confirmed PD/ death due to any cause or censoring whichever occurred first (maximum of 15 months);COTA:Initiation of first line post TCR MM to PD/ death due to any cause or censoring whichever occurred first (maximum of 64.3 months)
Population: Eligible participants whose data was retrieved and was used in this retrospective cohort study. Kaplan Meier method was used for analysis. Participants without an event were censored at the date of last adequate disease assessment or the data cut-off.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | C1071003 Cohort A | RWD: COTA
Number analyzed (Participants) | 123 | 239
Months | NA [NA to NA] — Median and 95% CI was not estimated because of insufficient number of participants with the event. | 4.70 [3.09 to 5.98]
Statistical Analysis 1: Comparison: C1071003 Cohort A vs RWD: COTA; Test type: Superiority; p < .0001, Regression, Cox; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.37 to 0.71] — Hazard ratios (HRs) were estimated using unadjusted Cox proportional hazard models

2. Primary Outcome: PFS: C1071003 Cohort A Versus COTA Cohort- Using Inverse Probability of Treatment Weights (IPTW)
Description: PFS: a) C1071003 Cohort A: time from the date of the first dose until confirmed PD per IMWG criteria or death due to any cause, whichever occurred first; b) COTA: time from initiation of the first line after participant identified as having TCR MM to either the date of progression or death due to any cause, whichever occurred first. IMWG criteria for progression: an increase of >=25% from the lowest response value in any 1 or more of the criteria: SPEP with an absolute increase >0.5 g/dL; 24-hour UPEP with an absolute increase >200 mg/24 h; in participants without measurable serum and urine M-protein, the absolute increase of >10 mg/dL in the difference between involved and uninvolved FLC levels; or an absolute bone marrow plasma cell percentage >10%. Retrospective data was retrieved and observed in the current study for approximately 1.5 months. Participants without an event were censored at date of last adequate disease assessment or the data cut-off. Kaplan Meier method was used.
Time Frame: as for outcome 1
Population: Eligible participants whose data was retrieved and was used in this retrospective cohort study. In this outcome measure, IPTW analysis was applied. IPTW eliminated the effect of confounding by observed baseline participant characteristics, improve covariate balance, and thereby obtained unbiased estimates of treatment effects. IPTW created pseudo-sets, hence "Number of Participants Analyzed" (N) are different from participant flow and baseline section.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | C1071003 Cohort A | RWD: COTA
Number analyzed (Participants) | 113 | 235
Months | NA [NA to NA] — Median and 95% CI was not estimated because of insufficient number of participants with the event. | 5.26 [3.25 to 6.28]
Statistical Analysis 1: Comparison: C1071003 Cohort A vs RWD: COTA; Test type: Superiority; p = .0003, Regression, Cox; Hazard Ratio (HR) = 0.37, 95% CI 2-sided [0.22 to 0.64] — IPTW HRs were estimated using weighted Cox proportional hazard models and confidence intervals were estimated using robust error variances

3. Primary Outcome: PFS: Study C1071003 Cohort A Versus Flatiron Cohort - Using Unweighted Analysis
Description: PFS: a) C1071003 Cohort A, PFS: time from the date of the first dose until confirmed PD per IMWG criteria or death due to any cause, whichever occurred first. B) Flatiron Health: time from initiation of the first line after participant identified as having TCR MM to either the date of progression or death due to any cause, whichever occurred first. IMWG criteria for progression: an increase of >= 25% from baseline/nadir value in any one or more of the following: an absolute increase in serum M-protein by SPEP by >= 0.5 g/dL; serum M-protein >= 1 g/dL if the lowest M component was >= 5 g/dL; an absolute increase in urine M-protein by UPEP by >=200 mg/24 h; in participants without measurable serum and urine M-protein levels, an absolute increase in the difference between involved and uninvolved FLC levels of >10 mg/dL. Retrospective data was retrieved and observed in the current study for approximately 1.5 months.
Time Frame: C1071003:First dose to confirmed PD/death due to any cause or censoring whichever occurred first(maximum of 15 months);Flatiron:Initiation of first line post TCR MM to PD/death due to any cause or censoring,whichever occurred first(maximum of 66.9 months)
Population: Eligible participants whose data was retrieved and was used in this retrospective cohort study. Kaplan Meier Method was used for analysis. Participants without an event were censored at date of last adequate disease assessment or the data cut-off.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | C1071003 Cohort A | RWD: Flatiron Health
Number analyzed (Participants) | 123 | 152
Months | NA [NA to NA] — Median and 95% CI was not estimated because of insufficient number of participants with the event. | 3.71 [3.02 to 7.13]

4. Primary Outcome: PFS: Study C1071003 Cohort A Versus Flatiron Cohort - Using IPTW Analysis
Description: PFS: a) C1071003 Cohort A, PFS: time from the date of the first dose until confirmed PD per IMWG criteria or death due to any cause, whichever occurred first. B) Flatiron Health: time from initiation of the first line after participant identified as having TCR MM to either the date of progression or death due to any cause, whichever occurred first. IMWG criteria for progression: an increase of >= 25% from baseline/nadir value in any one or more of the following: an absolute increase in serum M-protein by SPEP by >= 0.5 g/dL; serum M-protein >= 1 g/dL if the lowest M component was >= 5 g/dL; an absolute increase in urine M-protein by UPEP by >=200 mg/24 h; in participants without measurable serum and urine M-protein levels, an absolute increase in the difference between involved and uninvolved FLC levels of >10 mg/dL. Retrospective data was retrieved and observed in the current study for approximately 1.5 months. Kaplan Meier Method was used for analysis.
Time Frame: as for outcome 3
Population: Eligible participants whose data was retrieved and was used in this retrospective cohort study. IPTW analysis: eliminated the effect of confounding by observed baseline participant characteristics, improve covariate balance, and thereby obtained unbiased estimates of treatment effects. IPTW created pseudo-sets and "N" are different from participant and baseline section. Participants without an event were censored at date of last adequate disease assessment or the data cut-off.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | C1071003 Cohort A | RWD: Flatiron Health
Number analyzed (Participants) | 113 | 150
Months | NA [NA to NA] — Median and 95% CI was not estimated because of insufficient number of participants with the event. | 2.79 [1.87 to 5.59]

5. Secondary Outcome: Overall Survival (OS): Study C1071003 Cohort A Versus RWD COTA Cohort- Using Unweighted Analysis
Description: OS: a) C1071003 Cohort A: OS was defined as time from the date of the first dose until death due to any cause; b) COTA Cohort: OS was defined as time from initiation of the first line after participant identified as having TCR MM until the date of death due to any cause. Kaplan Meier Method was used for analysis. Participants without an event were censored at the latest available record or the data cut-off.
Time Frame: C1071003: The date of the first dose until death due to any cause or censoring (maximum up to 15 months); COTA: First line after participant identified as having TCR MM until the date of death due to any cause or censoring (maximum of 64.3 months)
Population: Eligible participants whose data was retrieved and was used in this retrospective cohort study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | C1071003 Cohort A | RWD: COTA
Number analyzed (Participants) | 123 | 239
Months | NA [NA to NA] — Median and 95% CI was not estimated because of insufficient number of participants with the event. | 11.24 [9.36 to 14.75]
Statistical Analysis 1: Comparison: C1071003 Cohort A vs RWD: COTA; Test type: Superiority; p = .0062, Regression, Cox; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.47 to 0.88] — HRs were estimated using unadjusted Cox proportional hazard models

6. Secondary Outcome: OS: Study C1071003 Cohort A Versus RWD COTA Cohort- Using IPTW Analysis
Description: as for outcome 5
Time Frame: as for outcome 5
Population: Eligible participants whose data was retrieved and was used in this retrospective cohort study. In this outcome measure, IPTW analysis was applied. IPTW eliminated the effect of confounding by observed baseline participant characteristics, improve covariate balance, and thereby obtained unbiased estimates of treatment effects. IPTW created pseudo-sets and "Number of Participants Analyzed" are different from participant flow and baseline section.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | C1071003 Cohort A | RWD: COTA
Number analyzed (Participants) | 113 | 235
Months | NA [NA to NA] — Median and 95% CI was not estimated because of insufficient number of participants with the event. | 11.24 [8.51 to 14.29]
Statistical Analysis 1: Comparison: C1071003 Cohort A vs RWD: COTA; Test type: Superiority; p = .0032, Regression, Cox; IPTW HRs were estimated using weighted Cox proportional hazard models and confidence intervals were estimated using robust error variances; Hazard Ratio (HR) = 0.46, 95% CI 2-sided [0.27 to 0.77]

7. Secondary Outcome: OS: Study C1071003 Cohort A Versus Flatiron Cohort - Using Unweighted Analysis
Description: OS: a) C1071003 Cohort A: OS was defined as time from the date of the first dose until death due to any cause; B) Flatiron Cohort: OS was defined as time from initiation of the first line after participant identified as having TCR MM until the date of death due to any cause. Kaplan Meier Method was used for analysis. Participants without an event were censored at the latest available record or the data cut-off.
Time Frame: C1071003: The date of the first dose until death due to any cause or censoring (maximum up to 15 months); Flatiron: First line after participant identified as having TCR MM until the date of death due to any cause or censoring (maximum of 66.9 months)
Population: Eligible participants whose data was retrieved and was used in this retrospective cohort study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | C1071003 Cohort A | RWD: Flatiron Health
Number analyzed (Participants) | 123 | 152
Months | NA [NA to NA] — Median and 95% CI was not estimated because of insufficient number of participants with the event. | 11.24 [7.75 to 13.21]

8. Secondary Outcome: OS: Study C1071003 Cohort A Versus Flatiron Cohort - Using IPTW Analysis
Description: as for outcome 7
Time Frame: as for outcome 7
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | C1071003 Cohort A | RWD: Flatiron Health
Number analyzed (Participants) | 113 | 150
Months | NA [NA to NA] — Median and 95% CI was not estimated because of insufficient number of participants with the event. | 11.24 [6.31 to 15.41]

ADVERSE EVENTS:
Time Frame: All-cause mortality: During observation period of approximately 15 months for C1071003, 64.3 months for RWD: COTA and 66.9 months for RWD: Flatiron Health; Serious adverse events and other adverse events: not applicable as adverse event data was not collected.
Description: This study is retrospective, it involves data that exist as structured data by the time of study start. From data source, individual participant data were not retrieved or validated. The minimum criteria for reporting an adverse event (AE) (i.e., identifiable participant, identifiable reporter, a suspect product, and event) cannot be met. Hence, adverse events were not planned to be collected and are not reported.
Arm/Group | C1071003 Cohort A | RWD: COTA | RWD: Flatiron Health
All-Cause Mortality (participants affected / at risk) | 55/123 | 171/239 | 90/152
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
IMWG: International Myeloma Working Group

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-05-15): https://cdn.clinicaltrials.gov/large-docs/90/NCT05932290/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-20): https://cdn.clinicaltrials.gov/large-docs/90/NCT05932290/SAP_001.pdf